CLINICAL TRIAL: NCT04238325
Title: Spanish Validation of the Frustration Discomfort Scale
Brief Title: Spanish Validation Frustration Discomfort Scale
Status: Completed | Type: Observational
Sponsor: Universitat Jaume I (Other)
Collaborators: Universidad de Zaragoza (Other); University of Seville (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Other Study IDs: FrustrationUJI
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: General Population, no Specific Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study aimed at validating the Frustration Discomfort Scale (Harrington, 2005). A back-translation process was followed to obtain a translated version of the scale, which was refined after a discussion with several clinicians.

DETAILED DESCRIPTION:
In the study, the Spanish adaptation of the Frustration Discomfort Scale will be disseminated with an online questionnaire using the Qualtrics platform. Additional questionnaires to explore the validity of the adapted scale will also be administered. Participants who complete the questionnaires and provide a valid ID number will enter a participate in a raffle to win an Amazon coupon of 40 euros. Ten coupons will be offered in total amongst participants.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Signs the informed consent
* Can read and understand Spanish
* Has access to a computer, a tablet or a smartphone with an internet connection

Exclusion Criteria:

* Being younger than 18 years of age
* Does not sign the informed consent
* Cannot read or understand Spanish
* Does not have access to a computer, a tablet or a smartphone with an internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This protocol will be disseminated globally to the population in Spain with no restriction. The maximum efforts will be made to disseminate the study to a wide range of individuals
Sampling Method: Probability Sample
Enrollment: 1513 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Frustration Discomfort Scale | The measure will be administered 1 day once only together with the remaining measures
  This is a measure of frustration intolerance. The original English version has been translated using a back-translation method and discussions about item have been made with clinicians with expertise in the field. The scale has 28 items that are gouped in 4 subscales. Items have a 1-to-5 response scale ranging from "nothing" to "a lot"

SECONDARY OUTCOMES:
Rosenberg self-esteem scale | The measure will be administered 1 day once only together with the remaining measures
  This scale of self-esteem has 10 items with responses ranging from 1 (completely agree) to 4 (completely disagree). This measure will be used for concurrent criterion validity analyses
Satisfaction with life scale | The measure will be administered 1 day once only together with the remaining measures
  This 5-item scale measures an individual's satisfaction with life using response options ranging from 1 (completely disagree) to 5 (completely agree). This measure will be used for concurrent criterion validity analyses
Acceptance and action questionnaire - II | The measure will be administered 1 day once only together with the remaining measures
  This 7-item scale measures acceptance of difficult experiences using a 7-point response scale (1= never true; 7=always true). This measure will be used for construct validity analyses
STAXI - 2 (trait anger scale only) | The measure will be administered 1 day once only together with the remaining measures
  The trait anger scale of the STAXI-2, which has 10 items, will be used to evaluate trait anger. The responses in the scale range from 1="not at all" to 4="very much". This measure will be used for concurrent criterion validity analyses
Irrational Procrastination Scale | The measure will be administered 1 day once only together with the remaining measures
  This 9-item scale will be administered to measure perceived procrastination. Items in the scale have a 5-point range (1=does not describe me at all; 5=decribes me completely). This measure will be used for concurrent criterion validity analyses
Trait Injustice Experiences Questionnare | The measure will be administered 1 day once only together with the remaining measures
  This measure of perceived trait injustice beliefs has 12 items, with responses ranging from 0="never" to 4="always". This measure will be used for construct validity analyses
European version of the Perceived Stress Scale | The measure will be administered 1 day once only together with the remaining measures
  This 10-item measure of perceived stress will be used for concurrent criterion validity analyses. Responses in the scale range from 0="never" to 4="very frequently"
Patient Health Questionnaire | The measure will be administered 1 day once only together with the remaining measures
  This 10-item measure of depressive symptoms will be used for concurrent criterion validity analyses. Response scales range from 0="None of the days" to 3="Almost all days"
General Anxiety Disorder scale | The measure will be administered 1 day once only together with the remaining measures
  This 7-item measure of anxiety symptoms will be used for concurrent criterion validity analyses. Response scales range from 0="None of the days" to 3="Almost all days"
General Attitudes and Beliefs Scale - reduced | The measure will be administered 1 day once only together with the remaining measures
  A shortened, 12-item version of the General Attitudes and Beliefs Scale will be administered. This measure will be used for concurrent criterion validity analyses. Responses in the scale have a 1-5 range (1="completely disagree"; 5="completely agree")

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psycholoy. Jaume I University, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No
Only the main PI will have access to the data.